CLINICAL TRIAL: NCT05360901
Title: A Pilot Study Aimed at Developing Automated Motivational Messaging for Patient Engagement With Digital Mental Health Interventions
Brief Title: Toward Understanding Drivers of Patient Engagement With Digital Mental Health Interventions - Part I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Jessica M. Lipschitz, Ph.D., Associate Director, BWH Digital Behavioral Health & Informatics Research Program, Brigham and Women's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020P000444; K23MH120324 (NIH)
Record Dates: First submitted 2022-04-29; First posted 2022-05-04 (Actual); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-11

CONDITIONS: Depression, Anxiety
Keywords: mHealth; Engagement; Depression; Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Single group, micro-randomized pilot trial design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IntelliCare with automated motivational messaging (Other): Digital mental health intervention with micro-randomized automated motivational messaging delivery
  Interventions: Behavioral: IntelliCare with automated motivational messaging

INTERVENTIONS:
Behavioral: IntelliCare with automated motivational messaging — Digital mental health intervention with automated motivational messaging

SUMMARY:
This pilot study is a precursor to a subsequent clinical trial that will test the impact of a set of automated motivational messages on patient engagement with a digital mental health intervention. The pilot study aims to systematically employ patient feedback to develop the automated motivational messages that will be used in the subsequent clinical trial.

DETAILED DESCRIPTION:
This is an in situ user-centered design pilot study to generate feedback on the automated motivational messaging the investigators are developing. Participants will download a digital mental health intervention (IntelliCare) to use for three weeks. During this three-week period, participants will receive automated motivational messages on a randomized schedule. That is, each day they will be randomized to either receive an automated motivational message (60% likelihood) or not receive an automated motivational message (40% likelihood). On days when a participant receives a message, the participant will be prompted to complete a brief survey on their reaction to the message received. At the end of three weeks, participants will be asked to complete a qualitative interview to provide further feedback on messages under development.

The primary outcome in this study is participant ratings from the brief surveys provided after automated motivational message delivery. We will also, however, look at participant feedback on messages under development in the qualitative interview as well as whether receiving a message makes users more likely to engage with the DMHI (IntelliCare) during the three hours following message delivery.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-80
* Patient Health Questionnaire-8 (PHQ-9) score≥10 and/or Generalized Anxiety Disorder-7 (GAD-7) Score≥8 indicating clinically significant depression or anxiety respectively
* Owns a smartphone
* Fluent in English
* Individual has a Mass General Brigham primary care provider

Exclusion Criteria:

* Diagnosis of bipolar disorder, any psychotic disorder, or a current substance use disorder per patient's report or medical record.
* Acute and/or unstable medical problem that may interfere with participation (e.g., scheduled for surgery in the next two months).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-07-06 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica M Lipschitz, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited via Massachusetts General Brigham Listservs and patient registries between June 2022 and September 2022. The first participant was enrolled on July 6, 2022 and the last participant was enrolled on September 22, 2022.
Period: Overall Study
Arm/Group | IntelliCare With Automated Motivational Messaging
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | IntelliCare With Automated Motivational Messaging
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.17 (14.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Generalized Anxiety Disorder-7 (GAD-7) [Mean (Standard Deviation); unit: units on a scale] — Generalized Anxiety Disorder-7 (GAD-7) is a self-report questionnaire used to screen for and measure the severity of anxiety disorders. Total scores range from 0-21, with higher scores indicating greater severity of anxiety symptoms.
  units on a scale | 13.33 (3.60)
Patient Health Questionnaire-8 (PHQ-8) [Mean (Standard Deviation); unit: units on a scale] — Patient Health Questionnaire-8 (PHQ-8) is a self-report questionnaire used to screen for and measure the severity of depression. Total scores range from 0-24, with higher scores indicating greater severity of depressive symptoms.
  units on a scale | 11.08 (5.98)

OUTCOME MEASURES:

1. Primary Outcome: Message Motivation Ratings
Description: Mean Likert scale rating of how well participants felt each message motivated them to use the digital mental health intervention as rated within 24 hours of message delivery. The Likert scale will range from 1 (not at all motivating) to 10 (very motivating) with a score of 5 being neutral.
Time Frame: 24 hours from message delivery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntelliCare With Automated Motivational Messaging
Number analyzed (Participants) | 12
units on a scale | 6.33 (2.02)

2. Secondary Outcome: Message Likability Ratings
Description: Mean Likert scale rating of how much participants liked each message as rated within 24 hours of message delivery. The Likert scale will range from 1 (hated the message) to 10 (loved the message) with a score of 5 being neutral.
Time Frame: 24 hours from message delivery
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | IntelliCare With Automated Motivational Messaging
Number analyzed (Participants) | 12
units on a scale | 6.35 (1.95)

3. Secondary Outcome: Engagement
Description: Percent of instances of message delivery that prompted user to launch the digital mental health intervention within 3 hours of delivery.
Time Frame: 3 hours from message delivery
Measure: Mean (Standard Deviation); unit: percent of messages resulting in app use
Arm/Group | IntelliCare With Automated Motivational Messaging
Number analyzed (Participants) | 12
percent of messages resulting in app use | 23.84 (21.51)

ADVERSE EVENTS:
Time Frame: 21 days
Arm/Group | IntelliCare With Automated Motivational Messaging
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-28): https://cdn.clinicaltrials.gov/large-docs/01/NCT05360901/Prot_SAP_000.pdf
  • Informed Consent Form (2022-08-08): https://cdn.clinicaltrials.gov/large-docs/01/NCT05360901/ICF_001.pdf